CLINICAL TRIAL: NCT02656576
Title: Detection of Human Papillomavirus in Polymerase Chain for Suspicious Lesions of the Amygdala: Concordance Smear-Biopsy
Acronym: HPV-BIOFRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10 153 02
Record Dates: First submitted 2015-11-02; First posted 2016-01-15 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Human Papillomavirus
Keywords: Human Papillomavirus; oropharynx biopsy; tonsillar lesion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patient with suspected lesions of the tonsillar region (Other): patients will have a tonsil biopsy and a smear
  Interventions: Procedure: Tonsil Biopsy; Procedure: Smear

INTERVENTIONS:
Procedure: Tonsil Biopsy — Biopsies were obtained during endoscopy of Aero-Digestive Tract Superior under general anesthesia.
Procedure: Smear — The smears are made in consultation a fortnight before performing endoscopic examination. They are carried out after a local anesthetic spray in order to optimize the number of cells collected.

SUMMARY:
Multicentre prospective study of concordance between two tissue sampling modes (smear / biopsy), which applies the same diagnostic method (PCR).

ELIGIBILITY:
Inclusion Criteria:

* Presents a suspicious lesion of the amygdala region
* Have a biopsy of the oropharynx planned in the operating room.

Exclusion Criteria:

* Pregnant Patient.
* Against anesthetic or surgical indication for endoscopy of the upper aerodigestive tract.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
the correlation between the two sampling methods | 1 month
  the correlation between the two sampling methods (smear and biopsy), defined by the probability of positive correlation and the negative concordance probability.

SECONDARY OUTCOMES:
rate of concordance for the detection of HPV between biopsy and smear | 1 month
the overall agreement | 1 month
  the overall agreement, assessed by kappa Cohen.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin VAIREL, Doctor, Principal Investigator — University Hospital, Toulouse
Locations (2):
- France (2):
  - CHU Toulouse, Toulouse
  - Institut Claudius Regaud, Toulouse